CLINICAL TRIAL: NCT06868537
Title: A Randomized Controlled Trial of the Launching! to Adulthood Program
Brief Title: A Trial of the Launching! to Adulthood Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Antonio Pagan, Postdoctoral Research Fellow II, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-25-0098
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Launching intervention
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Launching! to adulthood group therapy (Experimental)
  Interventions: Behavioral: Launching! to adulthood group therapy
- No intervention then Launching! to adulthood group therapy (Active Comparator)
  Interventions: Behavioral: Launching! to adulthood group therapy; Behavioral: standard of care

INTERVENTIONS:
Behavioral: Launching! to adulthood group therapy — Participants will be in a 12-week therapy program that includes weekly group sessions and individual coaching.
Behavioral: standard of care — Participants will receive a list of resources
  Arms: No intervention then Launching! to adulthood group therapy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Launching intervention (Pagan et al., 2024) in improving adaptive functioning, transition readiness, and social cognition in young adults with Autism Spectrum Disorder (ASD), compared to a delayed treatment control group, to examine whether the Launching intervention leads to improvements in executive functioning, co-occurring mental health symptoms, and quality of life, as measured by caregiver and self-report assessments, to assess the maintenance of treatment gains 12 weeks post-treatment and to replicate the findings of the Launching pilot study in an independent sample of young adults with ASD.

ELIGIBILITY:
Inclusion Criteria:

* confirmed case of ASD from a licensed mental health or medical professional
* score of >14 on the Social Communication Questionnaire-Lifetime (SCQ-L) completed with the mother or father
* meet DSM-5 criteria for ASD based on a Diagnostic and Statistical Manual of Mental Disorders (DSM-5) ASD symptom checklist
* willing and motivated to participate in the treatment
* a parent willing to participate
* verbal intelligence quotient (IQ) score >70 as assessed by the Kaufman Brief Intelligence Test 2nd edition revised (KBIT-2-R)

Exclusion Criteria:

* history of a psychotic disorder or current psychotic symptoms
* suicidal ideation with intent or plan
* current alcohol or other substance use disorder rated severe
* concurrent enrollment in another clinical trial for autism spectrum disorder
* expression of unwillingness to complete study procedures

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in adaptive functioning as assessed by the Adaptive Behavior Assessment System, Third Edition (ABAS-3) | Baseline, week 12, week 24
  This is a 239 item questionnaire and each is scored from 0(is not able to do this behavior) to 3 [(always able to do this behavior)(or almost always)] a higher number indicating better outcome
Change in social response as assessed by the Social Responsiveness Scale, Second Edition (SRS-2) | Baseline, week 12, week 24
  This is a 65 item questionnaire and each is scored on a 4-point Likert scale from 1(Not True) to 4(Almost Always True) for a maximum raw score of 120, higher score indicating worse outcome.
Change in transition readiness as assessed by the Transition Readiness Scale (TRS)-child version | Baseline, week 12, week 24
  This is a 30 item questionnaire and each is scored from 1(not true for me ) to 4(true for me) for a maximum score of 120, higher score indicating better outcome.
Change in transition readiness as assessed by the Transition Readiness Scale (TRS)-parent version | Baseline, week 12, week 24
  This is a 30 item questionnaire and each is scored from 1(not true for them) to 4(true for them) for a maximum score of 120, higher score indicating better outcome.

SECONDARY OUTCOMES:
Change in executive functioning as assessed by the Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) | Baseline, week 12, week 24
  This is a 75 item questionnaire and each is scored from 1(never) to 3(often) for a maximum score of 225, higher number indicating worse outcome
Change in depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) for depressive symptoms | Baseline, week 12, week 24
  This is a 9 item questionnaire and each is scored from 0(not at all) to 3(nearly every day) for a maximum score of 27, higher number indicating worse outcome
Change in anxiety as assessed by the Generalized Anxiety Disorder-7 (GAD-7) for anxiety symptoms | Baseline, week 12, week 24
  This is a 7 item questionnaire and each is scored from 0(not at all) to 4(nearly every day) for a maximum score of 21 , higher score indicating more anxiety
Change in quality of life as assessed by the World Health Organization Quality of Life Brief Version (WHOQOL-BREF) | Baseline, week 12, week 24
  This is a 26 item questionnaire ,with 4 domains. Each is scored from 1(very poor) to 5(very good) ,questions 3,4 and 26 are reverse scored for a maximum raw score of 120 and higher score indicating better quality of life
Change in quality of life as assessed by the Autism Spectrum Quality of Life (ASQoL) questionnaire | Baseline, week 12, week 24
  This is a 9 item questionnaire. Each is scored on a 4-point Likert scale from 1(not at all) to 5(totally) ,questions 6,7 and 8 are reverse scored for a maximum score range of 9-36 and higher score indicating better quality of life
Change in parental stress as assessed by the Parental Stress Scale (PSS) | Baseline, week 12, week 24
  This is a 14 item questionnaire and each item is scored from 1 (strongly disagree) to 5 (strongly agree) for a score range of 18-90, higher score indicating more stress

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pagan, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No